CLINICAL TRIAL: NCT05309148
Title: Investigation of the Effectiveness of Rehabilitation Equipment Based on Visual Feedback Technology (Eye Tracking) in Patients Who Have Suffered a Cerebral Stroke
Brief Title: Oculomotor and Cognitive Rehabilitation Using Visual Feedback in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Eye001
Record Dates: First submitted 2022-03-15; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Stroke; Oculomotor; Disorder; Attention Disturbances
Keywords: Eye tracking; Visual feedback; Cognitive functions; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training on eye tracker based device (Experimental): Patients will undergo a primary diagnostics of cognitive functions (memory, thinking skills, language, visual-spatial and communicative functions) and an diagnostics of the visual attention index on an eye tracker-based device. Based on the results of the diagnosis, participants will be offered a scheme of correctional training and secondary diagnostics at the end of training. Correctional training on an eye tracker-based device consists, firstly, of a 10-minute exercise at the beginning of each lesson aimed at improving visual functions and attention. Patients had to follow a spontaneously moving object. Secondly, correctional training includes a block of neurorehabilitation (simple cognitive exercises similar to the tasks presented in the assessment).
  Interventions: Behavioral: Training on eye tracker based device
- Training with a neuropsychologist (Active Comparator): Patients will undergo primary and secondary diagnostics on an eye tracker-based device, then participants will have a conventional correctional training with a neuropsychologist according to an individual correction plan.
  Interventions: Behavioral: Training with a neuropsychologist
- Training on eye tracker based device and with a neuropsychologist (Active Comparator): Patients will undergo primary and secondary diagnostics and correctional training on an eye tracker-based device, in the same time participants will have a conventional correctional training with a neuropsychologist according to an individual correction plan.
  Interventions: Behavioral: Training on eye tracker based device and with a neuropsychologist

INTERVENTIONS:
Behavioral: Training on eye tracker based device — The intervention is based on the principle of visual biofeedback. The patient sees where his gaze is and can objectively assess and correct his visual error.
  Arms: Training on eye tracker based device
Behavioral: Training with a neuropsychologist — The intervention is based on classical neuropsychological techniques aimed at correcting oculomotor disorders and improving visual attention (blank, psychometric, etc.)
  Arms: Training with a neuropsychologist
Behavioral: Training on eye tracker based device and with a neuropsychologist — This is combination of the first and second interventions
  Arms: Training on eye tracker based device and with a neuropsychologist

SUMMARY:
Investigators will test the effectiveness of oculomotor cognitive training using eye tracker-based device during rehabilitation course in patients with a degree of disability no more than 3 points on a scale Rankin.

DETAILED DESCRIPTION:
After a stroke, a wide range of neurological disorders can occur. One of them is impairments of the visual-oculomotor system in 8-31% of cases. Such patients experience loss of visual fields, hemianopia, tunnel vision, diplopia. All this causes great difficulties for returning to everyday life, as well as to professional activity. The eye tracking method allows to diagnose and evaluate the effectiveness of training aimed at improving the functioning of the saccadic system, reducing the volume of visual deficit. Currently, eye tracking is represented by a variety of technological solutions, but not all of them are used in the clinic.

The aim of the study is the application of an eye tracking-based device in cerebral stroke survivors for the correction of oculomotor disorders and visual attention functions.

Stroke patients participate in the study in Federal Center of Brain Research and Neurotechnologies of the Federal Medical Biological Agency, Moscow, Russia. The study has been conducted since January, 10 and was approved by a local ethic committee and followed principles of the Declaration of Helsinki. The patients stay in a 24-hour hospital and undergo a rehabilitation course. For 3 weeks, patients receive daily training on the C-Eye Pro device, AssisTech Sp. z. o. o, Poland. The patients interact with the device only by using eye movements. Participants undergo a primary assessment of cognitive functions (memory, thinking skills, language, visual-spatial and communicative functions). According to the results of the diagnosis, participants are offered a scheme of correctional training and secondary assessment at the end of the training. Correction training consists, firstly, of 10-minute exercise at the beginning of each session, aimed at improving visual functions and attention. Patients have to follow the spontaneously moving object. The result is evaluated qualitatively using heat and scanpath maps. Secondly, the correctional training includes a block of neurorehabilitation (simple cognitive exercises similar to the tasks presented in assessment).

ELIGIBILITY:
Inclusion Criteria:

* signed consent
* at least 3 points on the Rankin scale;
* the presence of disorders of the visual-oculomotor system, visual attention;
* understanding and following instructions; stable vegetative and hemodynamic parameters;
* on the MOOCA scale >22;
* patients should be fully examined for the underlying and concomitant disease (examination by a neurologist, ophthalmologist, physiotherapist);

Exclusion Criteria:

* 4, 5 points on the Rankin scale;
* unstable hemodynamics;
* time after stroke is less than 2 weeks;
* presence of epileptic activity;
* serious ophthalmological disorders (for example, partial atrophy of the optic nerve);

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Consciousness Test | Change from baseline at 2 weeks
  It is necessary to monitor the emerging stimuli (red circles) and keep eyes in the center of each of them. The quantitative indicator of visual attention as a percentage will be measured.
Cognitive function scale: memory scale | Change from baseline at 2 weeks
  Diagnostics of memory functions. Scale is evaluated as a percentage (min - 0%, max - 100%), the higher score means better performance
Cognitive function scale: language scale | Change from baseline at 2 weeks
  Diagnostics of language functions. Scale is evaluated as a percentage. (min - 0%, max - 100%), the higher score means better performance
Cognitive function scale: visual-spatial scale | Change from baseline at 2 weeks
  Diagnostics of visual-spatial functions. Scale is evaluated as a percentage. (min - 0%, max - 100%), the higher score means better performance
Cognitive function scale: communicative scale | Change from baseline at 2 weeks
  Diagnostics of communicative functions. Scale is evaluated as a percentage. (min - 0%, max - 100%), the higher score means better performance
Cognitive function scale: thinking skills scale | Change from baseline at 2 weeks
  Diagnostics of thinking skills functions. Scale is evaluated as a percentage. (min - 0%, max - 100%), the higher score means better performance
Assessment of a neuropsychologist | Change from baseline at 2 weeks
  Screening for cognitive impairment: MoCA (Montreal Cognitive Assessment), the results vary between 0 and 30 points. A score of 26 points or more is considered the norm. The lower the score, the worse the result
Assessment of a neuropsychologist | Change from baseline at 2 weeks
  Qualitative assessment of neuropsychological examination data (Luria-Nebraska neuropsychological battery)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Shurupova, Ph.D., Principal Investigator — Federal Center of Brain Research and Neurotechnologies of the Federal Medical Biological Agency
Locations (1):
- Federal Center of Brain Research and Neurotechnologies of the Federal Medical Biological Agency, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No